CLINICAL TRIAL: NCT06204718
Title: Preventing Pelvic Floor Dysfunction With Standard and Reflexive Pelvic Floor Exercises in Addition to Global Postural Re-education
Brief Title: Preventing Pelvic Floor Dysfunction With Pelvic Floor Exercises
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bandırma Onyedi Eylül University (Other)
Collaborators: Ebru Kaya Mutlu (Unknown)
Responsible Party: Principal Investigator, Gizem Türkmen, Principal Investigator, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-30
Record Dates: First submitted 2023-12-19; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Prevention Pelvic Muscle Dysfunction
Keywords: Global postural re-education; Reflexive Pelvic Floor Exercises; Prevention pelvic floor dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard pelvic floor exercises (Experimental): Standard pelvic floor exercises in addition to Global Postural Reeducation training
  Interventions: Other: Standard pelvic floor exercises
- Involuntary reflexive pelvic floor exercises (Experimental): Involuntary reflexive pelvic floor exercises in addition to Global Postural re-education training
  Interventions: Other: Involuntary reflexive pelvic floor exercises

INTERVENTIONS:
Other: Standard pelvic floor exercises — Pelvic floor muscle exercises will be given as 2 separate exercises including fast and slow contractions. For fast contractions, participants will be asked to contract their pelvic floor muscles strongly, hold them contracted for 5 seconds, and then relax them. For slow contractions, participants will be asked to gradually contract the pelvic floor muscles, hold them at maximum contraction for 5 seconds, and relax them gradually. Participants will be asked to perform 10 slow contractions after every 10 fast contractions. The aim is to train strength, coordination, endurance, and symmetry of pelvic floor muscles, motor learning and control, dynamic lumbopelvic stability, pelvic floor, and abdominal co-contraction. Every day, 10 fast, and 10 slow contractions with a total of 20 repetitions will be applied without changing the number by modifying the exercises every week. It will be applied for a total of 12 weeks.
  Arms: Standard pelvic floor exercises
Other: Involuntary reflexive pelvic floor exercises — Reflexive exercises (jump, squat jump, etc.) with 20 repetitions per day will be applied to the participants for 12 weeks with modifications every week.
  Arms: Involuntary reflexive pelvic floor exercises

SUMMARY:
Study participants will be randomised into 2 groups. Group 1: 1st assessment + 6 weeks of Global Postural Reeducation training plus standard pelvic floor exercises + 2nd assessment + 6 weeks of Global Postural Reeducation training plus standard pelvic floor exercises + 3rd assessment 2nd Group: 1st assessment + 6 weeks of Global Postural Reeducation training plus involuntary reflexive pelvic floor exercises + 2nd assessment + 6 weeks of Global Postural Reeducation training plus involuntary reflexive pelvic floor exercises + 3rd assessment

DETAILED DESCRIPTION:
Voluntary participants who agreed to participate in the study will be randomised into 2 groups of 36 people each (standard pelvic floor exercises and involuntary reflexive pelvic floor exercises) with the "Research Randomizer" programme (https://www.randomizer.org/). Group 1 (36 people) will receive Global Postural Reeducation training plus standard pelvic floor exercises for 12 weeks, 7 days a week (Total 84 sessions, 15 sessions face to face, 69 sessions home programme). Even numbers will be included in the 2nd group (36 people) and involuntary reflexive pelvic floor exercises will be given in addition to Global Postural Reeducation training for 12 weeks, 7 days a week (Total 84 sessions, 15 sessions face-to-face, 69 sessions home programme). In the study, detailed pelvic floor training will be given to both groups and the same assessments will be made on the pelvic floor muscles. After the initial assessments are completed, both groups will be given a total of 42 sessions of standard and involuntary reflexive pelvic floor exercises for 6 weeks (7 days a week). Participants in both groups will be evaluated at the end of 6 weeks and the remaining 6 weeks exercise programme will be given according to the arranged programme. At the end of the 12th week, the participants will be evaluated again.

Group 1: 1st assessment + 6 weeks of Global Postural Reeducation training plus standard pelvic floor exercises + 2nd assessment + 6 weeks of Global Postural Reeducation training plus standard pelvic floor exercises + 3rd assessment 2nd Group: 1st assessment + 6 weeks of Global Postural Reeducation training plus involuntary reflexive pelvic floor exercises + 2nd assessment + 6 weeks of Global Postural Reeducation training plus involuntary reflexive pelvic floor exercises + 3rd assessment

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being a desk worker between the ages of 18-65
* No pelvic floor dysfunction
* Being a woman

Exclusion Criteria:

* Systemic diseases such as hypertension and diabetes mellitus
* Presence of respiratory disease (asthma, COPD, etc...)
* Hormone replacement therapy
* History of neurogenic bladder
* Gynaecological cancer or collagen disease
* Breastfeeding
* Pregnancy
* Early postnatal period (less than one year)
* Pelvic organ prolapse (POP) or gynecological surgery
* Menopause
* Psychiatric comorbidities and/or cognitive impairment
* Impossibility of intra-vaginal physiotherapeutic examination due to untreated active or recurrent urinary infection, haematuria, or vaginal pain during physiotherapy assessment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic Floor Distress Inventory-PFDI-20 | Baseline
  The inventory consists of 3 sub-dimensions and contains 20 questions in total. The number of questions of each sub-dimension is indicated next to the name of that sub-dimension (For example; KRADE-8 contains 8 questions in total. The answer option of each question is divided into two as no and yes. Yes option is graded from Unimportant to Very. No=0, and the level of the answer of Yes corresponds to Insignificant=1, Less=1, Less=2, Moderate=3, Very=4 points. The score calculation system of the inventory is as follows; the average score of each sub-dimension is multiplied by 25. The number of points of 3 sub-dimensions is summed and a number between 0-300 points is obtained. The higher the score, the more serious the individual's problems are.
Pelvic Floor Distress Inventory-PFDI-20 | 6 Weeks Later
  The inventory consists of 3 sub-dimensions and contains 20 questions in total. The number of questions of each sub-dimension is indicated next to the name of that sub-dimension (For example; KRADE-8 contains 8 questions in total. The answer option of each question is divided into two as no and yes. Yes option is graded from Unimportant to Very. No=0, and the level of the answer of Yes corresponds to Insignificant=1, Less=1, Less=2, Moderate=3, Very=4 points. The score calculation system of the inventory is as follows; the average score of each sub-dimension is multiplied by 25. The number of points of 3 sub-dimensions is summed and a number between 0-300 points is obtained. The higher the score, the more serious the individual's problems are.
Pelvic Floor Distress Inventory-PFDI-20 | 12 Weeks Later
  The inventory consists of 3 sub-dimensions and contains 20 questions in total. The number of questions of each sub-dimension is indicated next to the name of that sub-dimension (For example; KRADE-8 contains 8 questions in total. The answer option of each question is divided into two as no and yes. Yes option is graded from Unimportant to Very. No=0, and the level of the answer of Yes corresponds to Insignificant=1, Less=1, Less=2, Moderate=3, Very=4 points. The score calculation system of the inventory is as follows; the average score of each sub-dimension is multiplied by 25. The number of points of 3 sub-dimensions is summed and a number between 0-300 points is obtained. The higher the score, the more serious the individual's problems are.
The female sexual function index (FSFI) | Baseline
  This scale assesses six dimensions of sexual function: sexual desire (first 2 questions), sexual arousal (questions 3-6), lubrication (questions 7-10), orgasm (questions 11-13), satisfaction (questions 14-16) and pain or discomfort (e.g. pain associated with vaginal penetration, questions 17-19). The highest total raw score that can be obtained in this scale is 95.0 and the lowest raw score is 4.0. Factor loadings used for scoring the whole scale were determined as 0.6 for sexual desire, 0.3 for sexual arousal and lubrication, 0.4 for orgasm, satisfaction and pain/discomfort. After multiplication by factor loadings, the highest score is 36.0 and the lowest score is 2.0. Total score >22.7 indicates normal sexual function and ≤ 22.7 indicates sexual dysfunction.
The female sexual function index (FSFI) | 6 Weeks Later
  This scale assesses six dimensions of sexual function: sexual desire (first 2 questions), sexual arousal (questions 3-6), lubrication (questions 7-10), orgasm (questions 11-13), satisfaction (questions 14-16) and pain or discomfort (e.g. pain associated with vaginal penetration, questions 17-19). The highest total raw score that can be obtained in this scale is 95.0 and the lowest raw score is 4.0. Factor loadings used for scoring the whole scale were determined as 0.6 for sexual desire, 0.3 for sexual arousal and lubrication, 0.4 for orgasm, satisfaction and pain/discomfort. After multiplication by factor loadings, the highest score is 36.0 and the lowest score is 2.0. Total score >22.7 indicates normal sexual function and ≤ 22.7 indicates sexual dysfunction.
The female sexual function index (FSFI) | 12 Weeks Later
  This scale assesses six dimensions of sexual function: sexual desire (first 2 questions), sexual arousal (questions 3-6), lubrication (questions 7-10), orgasm (questions 11-13), satisfaction (questions 14-16) and pain or discomfort (e.g. pain associated with vaginal penetration, questions 17-19). The highest total raw score that can be obtained in this scale is 95.0 and the lowest raw score is 4.0. Factor loadings used for scoring the whole scale were determined as 0.6 for sexual desire, 0.3 for sexual arousal and lubrication, 0.4 for orgasm, satisfaction and pain/discomfort. After multiplication by factor loadings, the highest score is 36.0 and the lowest score is 2.0. Total score >22.7 indicates normal sexual function and ≤ 22.7 indicates sexual dysfunction.
Global Pelvic Floor Bother Questionnaire | Baseline
  The scale consists of 9 questions in total. The questions were graded as "yes" or "no" (0) according to whether they had the complaint or not, and if they answered yes, how much the complaint bothered them was graded as "not at all" (1), "very little" (2), "a little" (3), "quite" (4), "very much" (5). Each question was given a score between 1 and 5. The scoring system gives the same weight to each question. The total score is between 0 and 45. For a score between 0 and 100, the total score is averaged and multiplied by 20. A high score indicates a high number of complaints.
Global Pelvic Floor Bother Questionnaire | 6 Weeks Later
  The scale consists of 9 questions in total. The questions were graded as "yes" or "no" (0) according to whether they had the complaint or not, and if they answered yes, how much the complaint bothered them was graded as "not at all" (1), "very little" (2), "a little" (3), "quite" (4), "very much" (5). Each question was given a score between 1 and 5. The scoring system gives the same weight to each question. The total score is between 0 and 45. For a score between 0 and 100, the total score is averaged and multiplied by 20. A high score indicates a high number of complaints.
Global Pelvic Floor Bother Questionnaire | 12 Weeks Later
  The scale consists of 9 questions in total. The questions were graded as "yes" or "no" (0) according to whether they had the complaint or not, and if they answered yes, how much the complaint bothered them was graded as "not at all" (1), "very little" (2), "a little" (3), "quite" (4), "very much" (5). Each question was given a score between 1 and 5. The scoring system gives the same weight to each question. The total score is between 0 and 45. For a score between 0 and 100, the total score is averaged and multiplied by 20. A high score indicates a high number of complaints.
Overactive Bladder Questionnaire (OAB-V8) | Baseline
  The OAB-V8 consists of the first 8 questions of the OAB-q and has been proposed as an overactive bladder screening and awareness test.
Overactive Bladder Questionnaire (OAB-V8) | 6 Weeks Later
  The OAB-V8 consists of the first 8 questions of the OAB-q and has been proposed as an overactive bladder screening and awareness test.
Overactive Bladder Questionnaire (OAB-V8) | 12 Weeks Later
  The OAB-V8 consists of the first 8 questions of the OAB-q and has been proposed as an overactive bladder screening and awareness test.
Pelvic Muscle Assessment | Baseline
  The PERFECT Scale can be used to assess voluntary contraction strength (P), endurance (E), slow-twitch muscle fibre performance (R), fast-twitch muscle fibre performance (F), pelvic floor muscle contraction pattern (E), transversus abdominus muscle cocontraction (C) and involuntary contraction in response to increased intra-abdominal pressure (T).
Pelvic Muscle Assessment | 6 Weeks Later
  The PERFECT Scale can be used to assess voluntary contraction strength (P), endurance (E), slow-twitch muscle fibre performance (R), fast-twitch muscle fibre performance (F), pelvic floor muscle contraction pattern (E), transversus abdominus muscle cocontraction (C) and involuntary contraction in response to increased intra-abdominal pressure (T).
Pelvic Muscle Assessment | 12 Weeks Later
  The PERFECT Scale can be used to assess voluntary contraction strength (P), endurance (E), slow-twitch muscle fibre performance (R), fast-twitch muscle fibre performance (F), pelvic floor muscle contraction pattern (E), transversus abdominus muscle cocontraction (C) and involuntary contraction in response to increased intra-abdominal pressure (T).

SECONDARY OUTCOMES:
Waist/ Hip Ratio | Baseline
  Waist-to-hip ratio (WHR) is the waist circumference divided by the hip circumference
Waist/ Hip Ratio | 6 Weeks Later
  Waist-to-hip ratio (WHR) is the waist circumference divided by the hip circumference
Waist/ Hip Ratio | 12 Weeks Later
  Waist-to-hip ratio (WHR) is the waist circumference divided by the hip circumference
Estimating body fat | Baseline
  This technique is based on the compression of the skin fold to measure the skin and the subcutaneous fat layer beneath it. To improve accuracy, multiple readings are taken in each body region and these readings are averaged and evaluated. The most common application is to measure skinfold thickness from three or four areas of the body and estimate the percentage of BF using prognostic equations.
Estimating body fat | 6 Weeks Later
  This technique is based on the compression of the skin fold to measure the skin and the subcutaneous fat layer beneath it. To improve accuracy, multiple readings are taken in each body region and these readings are averaged and evaluated. The most common application is to measure skinfold thickness from three or four areas of the body and estimate the percentage of BF using prognostic equations.
Estimating body fat | 12 Weeks Later
  This technique is based on the compression of the skin fold to measure the skin and the subcutaneous fat layer beneath it. To improve accuracy, multiple readings are taken in each body region and these readings are averaged and evaluated. The most common application is to measure skinfold thickness from three or four areas of the body and estimate the percentage of BF using prognostic equations.
ICIQ-SF: International Consultation on Incontinence Questionnaire-Short Form | Baseline
  The International Consultation on Incontinence Questionaire Short Form (ICIQ-SF), which has Turkish validity and reliability, will be used to question the type, frequency, amount and effects of urinary incontinence on daily life.
ICIQ-SF: International Consultation on Incontinence Questionnaire-Short Form | 6 Weeks Later
  The International Consultation on Incontinence Questionaire Short Form (ICIQ-SF), which has Turkish validity and reliability, will be used to question the type, frequency, amount and effects of urinary incontinence on daily life.
ICIQ-SF: International Consultation on Incontinence Questionnaire-Short Form | 12 Weeks Later
  The International Consultation on Incontinence Questionaire Short Form (ICIQ-SF), which has Turkish validity and reliability, will be used to question the type, frequency, amount and effects of urinary incontinence on daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Kaya Mutlu, Professor, PhD, Study Director — Bandırma Onyedi Eylül University
Locations (1):
- Bandırma Onyedi Eylül University, Bandırma, Balıkesir, Turkey (Türkiye)